CLINICAL TRIAL: NCT03119961
Title: Phase 1/2 Open Single-arm Monocentric Study Evaluating the Tolerance and Interest of Transient Opening of the Blood-Brain Barrier by Low Intensity Pulsed Ultrasound With the SONOCLOUD® Implantable Medical Device in Mild Alzheimer's Disease Patients (MMSE 20-26)
Brief Title: Blood Brain Barrier Opening in Alzheimer' Disease
Acronym: BOREAL1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CarThera (Industry); BPIfrance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150101; 2016-004145-82 (EudraCT Number); B2016-A01637-44 (Other: IDRCB)
Record Dates: First submitted 2017-02-27; First posted 2017-04-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2020-11

CONDITIONS: Alzheimer Disease
Keywords: Amyloid Amyloid Plaque; Tau Protein; Sonication
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SONOCLOUD® (Experimental): BBB opening by ultrasound
  Interventions: Device: SONOCLOUD®

INTERVENTIONS:
Device: SONOCLOUD® — BBB opening by ultrasound
  Other Names: BBB opening

SUMMARY:
In Alzheimer's disease (AD) an imbalance between the production and clearance of the ß-amyloid peptide is hypothesized as the driving event of the disease. The decreased clearance of Aß could be partly linked to a progressive dysfunction of the brain vasculature and of the blood brain barrier (BBB). Among many possible explanations for these failures of the multiple clinical trials evaluating innovative drugs in AD, one is the lack of target engagement, as none of these drugs is able to readily cross BBB. This barrier acts as a wall that actively and passively prevents the crossing of molecules between the blood and the brain parenchyma compartments. Only 0.3% of intravenously injected anti-Aß immunoglobulins reach the brain despite a half-life of 15-20 days. Low intensity Focal ultrasound associated to microbubble injection can open the BBB in a non invasive way. These openings are reversible in 2 hours to 2 days depending on the intensity of the ultrasound. Ultrasound opening of the BBB was initially used in a transgenic mouse model of AD to increase the brain delivery of an anti-Aß antibody. In this article, the Aß load was reduced in ultrasound treated brain region. Surprisingly it was then demonstrated that the simple opening of the BBB without any adjunct anti-Aß treatment was able to drive the same Aß clearance effects. This is probably linked to endogenous antibodies that are able to penetrate the brain parenchyma and target Aß plaques. Four opening sessions elicited positive promnesic effects in these mice. Our group conceived and developed a mean to easily, reproductively and innocuously open the BBB. A unique extra-dural ultrasound emitter (sonoCloud®) is surgically implanted in the skull under local anesthesia. It emits low intensity contact ultrasound (LICU) that are not deterred by bone and thus are able to open the BBB.Preclinical studies show the SonoCloud® device is safe and efficient as it allowed reproducible and repeatable opening of the BBB in rabbits, dogs and non human primates. Drugs up to 2000 Kilo Daltons (kDa) are able to cross the BBB to reach the brain parenchyma in which the concentration of Carboplatin was increased by 700% in the BBB opened region. No adverse event was evidenced both clinically, by EEG, Evoked potential, MRI, 18 Fluorodeoxyglucose (FDG) PET and histology in the primates after 7 bi-monthly sessions of LICU BBB opening. SonoCloud® and its external generator have been certified by the academic start-up CarThéra (APHP, UPMC). Our multidisciplinary skills (neurology, neurosurgery, neuroimaging, basic science departments in the same University hospital setting) and our previous experience of BBB opening in Man give us the unique opportunity to translate this procedure from neuro-oncology to AD which could 1) Have a positive effect on brain lesion load and symptoms by itself and 2) allow anti-AD (or more broadly, central nervous system) drugs to engage their targe

DETAILED DESCRIPTION:
Background:

Alzheimer's disease is the most prevalent neurodegenerative disease totalizing 33 million patients worldwide. If nothing is done to decrease the incidence of 1.8 Million patient/year, the prevalence will double in the next 20 years.

Physiopathologically, the amyloid cascade remains the predominant hypothesis. It states that an imbalance between the production and clearance of the ß-amyloid peptide is the driving event of the disease, leading to Tau hyperphosphorylation and accumulation in neurons as neurofibrillary tangles, neurodegeneration (synaptic and neuronal loss) and cognitive impairment. The decreased clearance of Aß could be partly linked to a progressive dysfunction of the brain vasculature and of the BBB.

New sets of diagnosis criteria for AD have been proposed to address the low specificity (70%) of the previous ones, that could be one of the causes of failure of previous clinical trials. Among these new criteria, cerebrospinal fluid (CSF) biomarkers and positon emission tomography (PET) with new ligands of amyloid plaques and more recently tau deposition are indicators of the underlying histopathology of the disease, and can also be used to evaluate early intervention efficacy as they are pathologic in the preclinical phase of AD, its prodromal phase.

the investigators aim to test an innovative BBB opening procedure that could drastically decrease AD patients' brain lesion load and alleviate their symptomatology.

Scientific/medical questions:

1) What is the tolerance of LICU and the SonoCloud® device in a population of patients with mild AD? 2) What are the physiopathological impact of LICU BBB opening in these patients as asserted by amyloid and 18FDG PET-MRI?

Objectives:

For the first phase I clinical trial in the world using LICU in AD to repeatedly open the BBB.

Primary objective: To evaluate the tolerance of the BBB opening session in 5 AD patients (Adverse event recording, cognitive and MRI evaluations).

Co-primary objective: To assess the impact of BBB opening on the hallmark lesions of AD (Aß & Tau) through PET-MRI imaging (decrease of the standardized uptake value ratio (SUVR) after vs. before treatment in the left supramarginal gyrus and left (treated) vs. right (untreated) supramarginal gyrus).

Secondary objective: increase cognitive performance in AD patients through the repeated opening of the BBB in the left supramarginal gyrus

Methods :

Ten patients suffering from mild AD will be included in the study.

Protocol :

Seven BBB opening session will be performed at a bi-monthly rate focusing on the left supramarginal gyrus, a cortical structure known to be affected by both amyloid and tau lesions early on during the evolution of the disease. All adverse events induced by surgery itself or by the LICU will be recorded. Amyloid ß and Tau lesion load will be evaluated benefiting from the PET-MRI that allows to clearly evaluate fine changes in SUVR taking into account loco-regional cortical specificity (cortical thickness). PET image analysis.

Mean Standard Uptake Values Ratios (SUVR) will be calculated with cerebellar gray matter activity as reference in volumes of interest. Voxel-wise uptake will then be divided by this reference value to get SUVR maps. PET images will be corrected for motion and partial volume effect thanks to simultaneous MRI acquisition. To analyze the longitudinal PET data, each follow-up T1-weighted MRI will be co-registered to the baseline MRI, and a within-subject template image will be calculated by averaging the coregistered T1-weighted images. This mean image will be used to calculate optimal transformation parameters to Montreal Neurological Institute (MNI) space. Next, baseline and follow-up PET images will be co-registered to the baseline MRI, spatially normalized to MNI using this optimal transformation, and scaled with cerebellar gray uptake. Individual percent annual changes maps will be then calculated. These maps will represent the voxel-wise calculation of percent metabolic change after BBB opening.

The investigators think that the clinical trial will be well tolerated by the patients as the rate of local adverse events is expected to be 1% since the SonoCloud device implantation is extra dural (without dura opening). The implantation is performed under local anaesthesia in an outclinic fashion.

Drawbacks and possible solution to overcome the problems :

Among expected drawback the investigators will have to be very vigilant for Amyloid related imaging anomalies (ARIAs) due to the sudden entry of endogenous antibodies in the brain parenchyma of patients with Aß and Tau prevalent lesions. If these ARIAs were to happen, an amendment of the protocol could be devised to add steroids, or reduce ultrasound intensity, or extend time during each opening session, or reduce number of BBB opening session, or in last use immunosuppressive drugs prior to the opening of the BBB.

This is the first study worldwide with the means to safely, repeatedly and reproductively open the BBB in AD, or more broadly, in any neurodegenerative disease. It is noteworthy to consider that it is only a phase I study aiming to demonstrate the feasibility of the technique in a mild form of AD. If this is the case and even in the absence of a positive effect on the lesions and symptoms it will then be possible to propose new projects aiming to associate these safe BBB opening to anti-AD drugs. In fact, this study could pave the way for further treatment venues of various neurodegenerative disease that share a brain accumulation of proteins that cannot be readily targeted in case of BBB integrity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 85 years old
* Alzheimer's disease, typical or atypical according to International Working Group-2 (IWG-2) criteria,

  * diagnosed on the basis of a cognitive assessment and an MRI, showing one of the three most frequent phenotypic presentations of the disease (hippocampal amnesia or logopenic aphasia or syndrome of posterior cortical atrophy)
  * certified by the CSF assay of biomarkers of the AD ratio PTau / Aβ> 0.11.
* Mild disease (MMSE 20-26) but presently pejorative outcome: relatively young subject (<80 years), "rapid" cognitive decline and high CSF tau rate (> 600pg / mL, for A diagnostic threshold of Alzheimer's disease of 450pg / mL). The evaluation of the pejorative evolution will be validated by the Committee of Experts of the Memory Center (IM2A at Pitié-Salpêtrière Hospital)
* Patients under stable Alzheimer's treatment for at least 3 months prior to entry into the study and in which no change is envisaged in the next months in order to avoid a loss of chance for the patient and to consider an aggravation at cessation of treatment as an adverse event due to the opening of the BBB.
* Affiliate or beneficiary of Affiliated to the French Health care system
* Patient and caregiver (undertaking to accompany the participant to the various necessary medico-surgical visits and spending at least 3 hours per day with the patient) having signed, free and informed consent.

Exclusion Criteria:

* Allergy to Gadolinium, Xylocaine or any contraindication to contrast products used for brain imaging, or to drugs used in perioperative procedures.
* Contraindications to SonoVue®

  * hypersensitivity to sulfur hexafluoride
  * recent acute coronary syndrome or unstable ischemic heart disease
  * heart failure, chronic or acute stage III or IV,
  * patient undergoing drug therapy incorporating dobutamine,
  * severe pulmonary arterial hypertension
  * uncontrolled systemic hypertension,
  * respiratory distress syndrome
* Severe renal impairment with glomerular filtration rate (GFR) <30 mL / min / 1.73 m2 (Gadolinium IC)
* Hepatic impairment characterized by international normalized ratio (INR)> 1.5 or Factor V <50% of the standard.
* Patient taking an associated treatment considered potentially toxic to the central nervous system (CNS).
* Patient included or having participated in the 5 years preceding the inclusion in this study in another research protocol on Alzheimer's (medical treatment or medical device).
* Epilepsy or potentially pro-convulsive medication
* Ischemic or haemorrhagic stroke consisting of supracentimetric vascular leucopathy with a grade greater than 2 in the classification of Fazekas and Schmidt
* Presence of at least one lobar micro-bleeding identified in MRI performed in current care prior to inclusion (SWI sequence) in the sonication zone (left supramarginal gyrus)
* Chronic and abusive consumption of toxic (alcohol or drugs) except tobacco.
* Contra-indication to MRI (intracorporeal metallic material, claustrophobia)
* Hemostasis disorders (thrombocytopenia <75,000, prothrombin ratio (PR) <60%, INR> 1.5, antiplatelet therapy or anticoagulant in progress)
* Phlebitis or active pulmonary embolism
* Patient unable to perform cognitive tests (less than 7 years of study, mother tongue different from French, severe unpaired sensory disorder).
* Patient under judicial protection
* Absence of accompanying person
* Patient with an ongoing infection clinically characterized by febrile syndrome and possible calling points (cough, pain, skin lesion, etc.) OR biologically suspected on C-reactive protein(CRP)> 10, Procalcitonin> 0.1, positive examination of the urine (CBEU).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Florbetapir SUVr and Fluorodeoxyglucose MUV changes in BBB opening region of interest (ROI) | Change from baseline at 4month and 8 month
  PET MRI evaluation

SECONDARY OUTCOMES:
Adverse events recording | up to 9 months
  Clinical and MRI evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Stephane EPELBAUM, MD, PhD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- APHP - Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carpentier A, Canney M, Vignot A, Reina V, Beccaria K, Horodyckid C, Karachi C, Leclercq D, Lafon C, Chapelon JY, Capelle L, Cornu P, Sanson M, Hoang-Xuan K, Delattre JY, Idbaih A. Clinical trial of blood-brain barrier disruption by pulsed ultrasound. Sci Transl Med. 2016 Jun 15;8(343):343re2. doi: 10.1126/scitranslmed.aaf6086. PMID 27306666
- [Background] Horodyckid C, Canney M, Vignot A, Boisgard R, Drier A, Huberfeld G, Francois C, Prigent A, Santin MD, Adam C, Willer JC, Lafon C, Chapelon JY, Carpentier A. Safe long-term repeated disruption of the blood-brain barrier using an implantable ultrasound device: a multiparametric study in a primate model. J Neurosurg. 2017 Apr;126(4):1351-1361. doi: 10.3171/2016.3.JNS151635. Epub 2016 Jun 10. PMID 27285538
- [Background] Goldwirt L, Canney M, Horodyckid C, Poupon J, Mourah S, Vignot A, Chapelon JY, Carpentier A. Enhanced brain distribution of carboplatin in a primate model after blood-brain barrier disruption using an implantable ultrasound device. Cancer Chemother Pharmacol. 2016 Jan;77(1):211-6. doi: 10.1007/s00280-015-2930-5. Epub 2015 Dec 8. PMID 26645405
- [Background] Beccaria K, Canney M, Goldwirt L, Fernandez C, Piquet J, Perier MC, Lafon C, Chapelon JY, Carpentier A. Ultrasound-induced opening of the blood-brain barrier to enhance temozolomide and irinotecan delivery: an experimental study in rabbits. J Neurosurg. 2016 Jun;124(6):1602-10. doi: 10.3171/2015.4.JNS142893. Epub 2015 Nov 13. PMID 26566207
- [Background] Beccaria K, Canney M, Goldwirt L, Fernandez C, Adam C, Piquet J, Autret G, Clement O, Lafon C, Chapelon JY, Carpentier A. Opening of the blood-brain barrier with an unfocused ultrasound device in rabbits. J Neurosurg. 2013 Oct;119(4):887-98. doi: 10.3171/2013.5.JNS122374. Epub 2013 Jun 21. PMID 23790118
- [Background] Jordao JF, Ayala-Grosso CA, Markham K, Huang Y, Chopra R, McLaurin J, Hynynen K, Aubert I. Antibodies targeted to the brain with image-guided focused ultrasound reduces amyloid-beta plaque load in the TgCRND8 mouse model of Alzheimer's disease. PLoS One. 2010 May 11;5(5):e10549. doi: 10.1371/journal.pone.0010549. PMID 20485502
- [Background] Jordao JF, Thevenot E, Markham-Coultes K, Scarcelli T, Weng YQ, Xhima K, O'Reilly M, Huang Y, McLaurin J, Hynynen K, Aubert I. Amyloid-beta plaque reduction, endogenous antibody delivery and glial activation by brain-targeted, transcranial focused ultrasound. Exp Neurol. 2013 Oct;248:16-29. doi: 10.1016/j.expneurol.2013.05.008. Epub 2013 May 21. PMID 23707300
- [Background] Goldwirt L, Beccaria K, Carpentier A, Farinotti R, Fernandez C. Irinotecan and temozolomide brain distribution: a focus on ABCB1. Cancer Chemother Pharmacol. 2014 Jul;74(1):185-93. doi: 10.1007/s00280-014-2490-0. Epub 2014 May 28. PMID 24867782
- [Background] Goldwirt L, Beccaria K, Carpentier A, Idbaih A, Schmitt C, Levasseur C, Labussiere M, Milane A, Farinotti R, Fernandez C. Preclinical impact of bevacizumab on brain and tumor distribution of irinotecan and temozolomide. J Neurooncol. 2015 Apr;122(2):273-81. doi: 10.1007/s11060-015-1717-1. Epub 2015 Jan 13. PMID 25794638
- [Background] Helmer C, Peres K, Letenneur L, Guttierez-Robledo LM, Ramaroson H, Barberger-Gateau P, Fabrigoule C, Orgogozo JM, Dartigues JF. Dementia in subjects aged 75 years or over within the PAQUID cohort: prevalence and burden by severity. Dement Geriatr Cogn Disord. 2006;22(1):87-94. doi: 10.1159/000093459. Epub 2006 May 18. PMID 16710088
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Hardy J, Selkoe DJ. The amyloid hypothesis of Alzheimer's disease: progress and problems on the road to therapeutics. Science. 2002 Jul 19;297(5580):353-6. doi: 10.1126/science.1072994. PMID 12130773
- [Background] Hardy JA, Higgins GA. Alzheimer's disease: the amyloid cascade hypothesis. Science. 1992 Apr 10;256(5054):184-5. doi: 10.1126/science.1566067. No abstract available.
- [Background] Zlokovic BV. The blood-brain barrier in health and chronic neurodegenerative disorders. Neuron. 2008 Jan 24;57(2):178-201. doi: 10.1016/j.neuron.2008.01.003. PMID 18215617
- [Background] Dubois B, Feldman HH, Jacova C, Dekosky ST, Barberger-Gateau P, Cummings J, Delacourte A, Galasko D, Gauthier S, Jicha G, Meguro K, O'brien J, Pasquier F, Robert P, Rossor M, Salloway S, Stern Y, Visser PJ, Scheltens P. Research criteria for the diagnosis of Alzheimer's disease: revising the NINCDS-ADRDA criteria. Lancet Neurol. 2007 Aug;6(8):734-46. doi: 10.1016/S1474-4422(07)70178-3. PMID 17616482
- [Background] Dubois B, Feldman HH, Jacova C, Hampel H, Molinuevo JL, Blennow K, DeKosky ST, Gauthier S, Selkoe D, Bateman R, Cappa S, Crutch S, Engelborghs S, Frisoni GB, Fox NC, Galasko D, Habert MO, Jicha GA, Nordberg A, Pasquier F, Rabinovici G, Robert P, Rowe C, Salloway S, Sarazin M, Epelbaum S, de Souza LC, Vellas B, Visser PJ, Schneider L, Stern Y, Scheltens P, Cummings JL. Advancing research diagnostic criteria for Alzheimer's disease: the IWG-2 criteria. Lancet Neurol. 2014 Jun;13(6):614-29. doi: 10.1016/S1474-4422(14)70090-0. PMID 24849862
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Salloway S, Sperling R, Fox NC, Blennow K, Klunk W, Raskind M, Sabbagh M, Honig LS, Porsteinsson AP, Ferris S, Reichert M, Ketter N, Nejadnik B, Guenzler V, Miloslavsky M, Wang D, Lu Y, Lull J, Tudor IC, Liu E, Grundman M, Yuen E, Black R, Brashear HR; Bapineuzumab 301 and 302 Clinical Trial Investigators. Two phase 3 trials of bapineuzumab in mild-to-moderate Alzheimer's disease. N Engl J Med. 2014 Jan 23;370(4):322-33. doi: 10.1056/NEJMoa1304839. PMID 24450891
- [Background] Tapiola T, Alafuzoff I, Herukka SK, Parkkinen L, Hartikainen P, Soininen H, Pirttila T. Cerebrospinal fluid beta-amyloid 42 and tau proteins as biomarkers of Alzheimer-type pathologic changes in the brain. Arch Neurol. 2009 Mar;66(3):382-9. doi: 10.1001/archneurol.2008.596. PMID 19273758
- [Background] Clark CM, Schneider JA, Bedell BJ, Beach TG, Bilker WB, Mintun MA, Pontecorvo MJ, Hefti F, Carpenter AP, Flitter ML, Krautkramer MJ, Kung HF, Coleman RE, Doraiswamy PM, Fleisher AS, Sabbagh MN, Sadowsky CH, Reiman EP, Zehntner SP, Skovronsky DM; AV45-A07 Study Group. Use of florbetapir-PET for imaging beta-amyloid pathology. JAMA. 2011 Jan 19;305(3):275-83. doi: 10.1001/jama.2010.2008. PMID 21245183
- [Background] Klunk WE, Engler H, Nordberg A, Wang Y, Blomqvist G, Holt DP, Bergstrom M, Savitcheva I, Huang GF, Estrada S, Ausen B, Debnath ML, Barletta J, Price JC, Sandell J, Lopresti BJ, Wall A, Koivisto P, Antoni G, Mathis CA, Langstrom B. Imaging brain amyloid in Alzheimer's disease with Pittsburgh Compound-B. Ann Neurol. 2004 Mar;55(3):306-19. doi: 10.1002/ana.20009. PMID 14991808
- [Background] Rinne JO, Wong DF, Wolk DA, Leinonen V, Arnold SE, Buckley C, Smith A, McLain R, Sherwin PF, Farrar G, Kailajarvi M, Grachev ID. [(18)F]Flutemetamol PET imaging and cortical biopsy histopathology for fibrillar amyloid beta detection in living subjects with normal pressure hydrocephalus: pooled analysis of four studies. Acta Neuropathol. 2012 Dec;124(6):833-45. doi: 10.1007/s00401-012-1051-z. Epub 2012 Oct 10. PMID 23053137
- [Background] Chien DT, Bahri S, Szardenings AK, Walsh JC, Mu F, Su MY, Shankle WR, Elizarov A, Kolb HC. Early clinical PET imaging results with the novel PHF-tau radioligand [F-18]-T807. J Alzheimers Dis. 2013;34(2):457-68. doi: 10.3233/JAD-122059. PMID 23234879
- [Background] Shah M, Catafau AM. Molecular Imaging Insights into Neurodegeneration: Focus on Tau PET Radiotracers. J Nucl Med. 2014 Jun;55(6):871-4. doi: 10.2967/jnumed.113.136069. Epub 2014 May 15. PMID 24833492
- [Background] Zhang W, Arteaga J, Cashion DK, Chen G, Gangadharmath U, Gomez LF, Kasi D, Lam C, Liang Q, Liu C, Mocharla VP, Mu F, Sinha A, Szardenings AK, Wang E, Walsh JC, Xia C, Yu C, Zhao T, Kolb HC. A highly selective and specific PET tracer for imaging of tau pathologies. J Alzheimers Dis. 2012;31(3):601-12. doi: 10.3233/JAD-2012-120712. PMID 22683529
- [Background] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Background] Ossenkoppele R, Jansen WJ, Rabinovici GD, Knol DL, van der Flier WM, van Berckel BN, Scheltens P, Visser PJ; Amyloid PET Study Group; Verfaillie SC, Zwan MD, Adriaanse SM, Lammertsma AA, Barkhof F, Jagust WJ, Miller BL, Rosen HJ, Landau SM, Villemagne VL, Rowe CC, Lee DY, Na DL, Seo SW, Sarazin M, Roe CM, Sabri O, Barthel H, Koglin N, Hodges J, Leyton CE, Vandenberghe R, van Laere K, Drzezga A, Forster S, Grimmer T, Sanchez-Juan P, Carril JM, Mok V, Camus V, Klunk WE, Cohen AD, Meyer PT, Hellwig S, Newberg A, Frederiksen KS, Fleisher AS, Mintun MA, Wolk DA, Nordberg A, Rinne JO, Chetelat G, Lleo A, Blesa R, Fortea J, Madsen K, Rodrigue KM, Brooks DJ. Prevalence of amyloid PET positivity in dementia syndromes: a meta-analysis. JAMA. 2015 May 19;313(19):1939-49. doi: 10.1001/jama.2015.4669. PMID 25988463
- [Background] Doody RS, Thomas RG, Farlow M, Iwatsubo T, Vellas B, Joffe S, Kieburtz K, Raman R, Sun X, Aisen PS, Siemers E, Liu-Seifert H, Mohs R; Alzheimer's Disease Cooperative Study Steering Committee; Solanezumab Study Group. Phase 3 trials of solanezumab for mild-to-moderate Alzheimer's disease. N Engl J Med. 2014 Jan 23;370(4):311-21. doi: 10.1056/NEJMoa1312889. PMID 24450890
- [Background] Duits FH, Teunissen CE, Bouwman FH, Visser PJ, Mattsson N, Zetterberg H, Blennow K, Hansson O, Minthon L, Andreasen N, Marcusson J, Wallin A, Rikkert MO, Tsolaki M, Parnetti L, Herukka SK, Hampel H, De Leon MJ, Schroder J, Aarsland D, Blankenstein MA, Scheltens P, van der Flier WM. The cerebrospinal fluid "Alzheimer profile": easily said, but what does it mean? Alzheimers Dement. 2014 Nov;10(6):713-723.e2. doi: 10.1016/j.jalz.2013.12.023. Epub 2014 Apr 8. PMID 24721526
- [Background] Schindowski K, Bretteville A, Leroy K, Begard S, Brion JP, Hamdane M, Buee L. Alzheimer's disease-like tau neuropathology leads to memory deficits and loss of functional synapses in a novel mutated tau transgenic mouse without any motor deficits. Am J Pathol. 2006 Aug;169(2):599-616. doi: 10.2353/ajpath.2006.060002. PMID 16877359
- [Result] Epelbaum S, Burgos N, Canney M, Matthews D, Houot M, Santin MD, Desseaux C, Bouchoux G, Stroer S, Martin C, Habert MO, Levy M, Bah A, Martin K, Delatour B, Riche M, Dubois B, Belin L, Carpentier A. Pilot study of repeated blood-brain barrier disruption in patients with mild Alzheimer's disease with an implantable ultrasound device. Alzheimers Res Ther. 2022 Mar 8;14(1):40. doi: 10.1186/s13195-022-00981-1. PMID 35260178
- [Derived] Mathew AS, Gorick CM, Price RJ. Multiple regression analysis of a comprehensive transcriptomic data assembly elucidates mechanically- and biochemically-driven responses to focused ultrasound blood-brain barrier disruption. Theranostics. 2021 Oct 11;11(20):9847-9858. doi: 10.7150/thno.65064. eCollection 2021. PMID 34815790
- See also: Related Info — http://www.aphp.fr
- See also: Related Info — http://www.carthera.eu